CLINICAL TRIAL: NCT02803567
Title: Trial of a Novel Brief Intervention on Health Behaviors for Youth With Chronic Medical
Brief Title: Trial of a Novel Brief Intervention on Health Behaviors for Youth With Chronic Medical Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Conrad N. Hilton Foundation (Other)
Responsible Party: Principal Investigator, Sharon Levy, Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P00021649
Record Dates: First submitted 2016-03-03; First posted 2016-06-17 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Those in the intervention arm will receive a computerized brief intervention composed of tailored feedback and psycho-education on substance use. Content in the intervention will focus on health promotion and will deliver positive messages about health.
  Interventions: Behavioral: Brief psycho-educational intervention
- Control (No Intervention): Those in the control arm will receive treatment as usual.

INTERVENTIONS:
Behavioral: Brief psycho-educational intervention — Participants in the intervention arm will receive a computerized brief intervention composed of tailored feedback and psycho-education specific to their chronic condition.
  Arms: Intervention

SUMMARY:
The primary goal of this project is to develop a tailored screening, brief intervention and referral to treatment (SBIRT) model for youth with chronic medical conditions (YCMC) for delivery at point of care during a routine healthcare visit, through conducting a rigorous randomized control trial among adolescent patients with type 1 diabetes (TID) or rheumatologic conditions. The secondary goal is to assess the attitudes and knowledge of parents of these same adolescents, to explore links between parent beliefs and adolescent behavior around substance use.

DETAILED DESCRIPTION:
The proposed project is a randomized control trial to assess the efficacy of an SBIRT model tailored to youth with chronic medical conditions. This trial is being built into a larger, longitudinal cohort study to assess whether a set of brief, substance specific questions can accurately predict adolescent substance use outcomes when compared to more lengthy, criterion standard assessment questions, in cross-sectional and prospective analysis. The first component of the project will consist of pre-testing an assessment battery and brief electronic intervention with a small sample of 14-17 year old youth. In the second component the investigators will randomize consented eligible participants into intervention or control arms of the study and administer the 1) Baseline Assessment Battery and the 2) Brief Intervention OR Treatment as Usual (TAU). In the third component the investigators will follow up with all participants at 6 and then 12 months after study entry to reassess rates of substance use through follow up assessment batteries.

At baseline, the investigators will also attempt to enroll parents of all participants who are present at the time of enrollment. The investigators will separately consent and administer a brief assessment battery to parents to assess their knowledge and attitudes around substance use, as well as opinions and attitudes regarding other health and risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 year-old youth presenting for routine medical care in the Rheumatology clinic or Endocrinology clinic at Boston Children's Hospital (BCH)
* A diagnosis of type 1 diabetes for at least a year or a diagnosis of a Rheumatologic condition for at least a year.
* Able to read and understand English at a middle school level or greater
* Consent to participation in the study and consent to the 6 month and 12 month follow up assessments.

Exclusion Criteria:

* Patients who are medically or emotionally unstable or otherwise unable to provide assent at the time of their appointment as determined by their clinician or the research team
* Unable to speak/read English at a middle school reading level
* Unable to use a computer keyboard and/or complete an interviewer-assisted questionnaire
* Do not consent to 6 month and 12 month re-assessment.
* Patients who are pregnant at baseline

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 460 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Frequency and quantity of alcohol use in the past 12 months, measured using the Screen to Brief Intervention (S2BI) screening tool. | 12 months post intervention
  We will compare changes in frequency and quantity of alcohol use over the past twelve months between the intervention and treatment as usual groups.

SECONDARY OUTCOMES:
Frequency of marijuana use in the past 12 months, measured using the S2BI Screening Tool. | 12 months post intervention
  We will compare changes frequency of marijuana use in the past 12 months between the intervention and treatment as usual groups.
Perceived risk of harm of substance use | 12 months post intervention
  We will compare self-reported perceived risk of harm of substance use between intervention and TAU groups using Monitoring the Future questions.
Medication Adherence measured by self-report | 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, MPH, Principal Investigator — Boston Children's Hospital; Elissa Weitzman, ScD, MSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available. We will provide our findings in aggregate.

REFERENCES:
- [Derived] Weitzman ER, Minegishi M, Dedeoglu F, Fishman LN, Garvey KC, Wisk LE, Levy S. Disease-Tailored Brief Intervention for Alcohol Use Among Youths With Chronic Medical Conditions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2419858. doi: 10.1001/jamanetworkopen.2024.19858. PMID 38985475